CLINICAL TRIAL: NCT04630522
Title: A Randomized, Open-Label, Dose-finding, Multi-centre, Phase Ib Study toEvaluate the Efficacy and Safety of JMT103 in Patients With Bone Metastases From Solid Tumors
Brief Title: Efficacy and Safety of JMT103 in Patients With Bone Metastases From Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT103CN01-1
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Bone Metastases From Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMT103- 120 mg SC Q4W (Experimental): Eligible patients will receive JMT103 120 mg SC Q4W for up to 13 cycles.
  Interventions: Drug: Drug: JMT103- 120 mg SC Q4W; Dietary Supplement: Dietary Supplement: Calcium Dietary Supplement: Vitamin D
- JMT103- 120 mg SC Q8W (Experimental): Eligible patients will receive JMT103 120 mg SC Q8W for up to 7 cycles.
  Interventions: Drug: Drug: JMT103- 120 mg SC Q8W; Dietary Supplement: Dietary Supplement: Calcium Dietary Supplement: Vitamin D
- JMT103- 180 mg SC Q8W (Experimental): Eligible patients will receive JMT103 180 mg SC Q8W for up to 7 cycles.
  Interventions: Drug: Drug: JMT103- 180 mg SC Q8W; Dietary Supplement: Dietary Supplement: Calcium Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Drug: JMT103- 120 mg SC Q4W — JMT103 is administered subcutaneously at a dose of 120 mg on day 1 of each 4-week cycle.
  Arms: JMT103- 120 mg SC Q4W
Drug: Drug: JMT103- 120 mg SC Q8W — JMT103 is administered subcutaneously at a dose of 120 mg on day 1 of each 8-week cycle.
  Arms: JMT103- 120 mg SC Q8W
Drug: Drug: JMT103- 180 mg SC Q8W — JMT103 is administered subcutaneously at a dose of 180 mg on day 1 of each 8-week cycle.
  Arms: JMT103- 180 mg SC Q8W
Dietary Supplement: Dietary Supplement: Calcium Dietary Supplement: Vitamin D — Calcium is given orally at a dose of 500 mg at least, once daily. Vitamin D is given orally at a dose of 400 IU at least, once daily.

SUMMARY:
This is a randomized, open-label, dose-finding, multi-centre, phase Ⅰb study to evaluate the efficacy and safety of JMT103 in patients with bone metastases from solid tumors.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the efficacy and safety of JMT103 in patients with bone metastases from solid tumors.

Eligible patients will be randomly assigned to receive JMT103 120mg subcutaneously (SC) every 4 weeks (Q4W), 120mg subcutaneously (SC) every 8 weeks (Q8W) and 180mg subcutaneously (SC) every 8 weeks (Q8W) in a 1:1:1 ratio. Patients will receive the treatment until the completion of 48 weeks of treatment, intolerable toxicity, loss to follow-up, withdrawal (patient's decision or investigator's decision), whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and signed informed consent.
2. Male or female, 18 years and older.
3. Histologically/cytologically confirmed malignant solid tumors.
4. Radiographic evidence of at least one bone metastasis.
5. Eligible fertile patients (male and female) must agree to use an effective method of contraception with their partners from the signing of informed consent until at least 6 months after the last treatment.
6. Adequate organ functions.
7. Albumin-corrected serum calcium ≥ 1 x lower limit of normal (LLN) at screening (calcium supplement is not allowed within 8 hours prior to screening).
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
9. Life expectancy ≥ 6 months

Exclusion Criteria:

1. Previous or present osteomyelitis or osteonecrosis of the jaw; unhealed dental or oral surgery wounds; acute disease of the tooth or jaw requiring oral surgery; and invasive dental surgery planned to be received during the study;
2. Radiotherapy or orthopaedic surgery is planned for patients during the study;
3. Known symptomatic brain metastases.
4. Abnormal bone metabolism (such as Paget's disease, Cushing's syndrome, hyperprolactinemia), rheumatoid arthritis, parathyroid disease
5. Clinically significant disease (such as uncontrolled diabetes, congestive heart failure, hypertension>150/90 mmHg).
6. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection.
7. Systemic therapy of active bacterial infection or fungal infection within 7 days prior to randomization.
8. Pregnant or lactating women.
9. Prior use of antibody against nuclear factor kappa-B (NFκB) ligand (RANKL).
10. Participated in other clinical studies and received other experimental drugs within 4 weeks prior to randomization.
11. Prior use of bisphosphonate within 4 weeks prior to randomization.
12. Prior use of one of following osteoporosis medications within 6 months prior to randomization (Parathyroid hormone (PTH) analogue, calcitonin, osteoprotegerin, mithramycin, and strontium).
13. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for the toxicity without safety risk judged by the investigator, such as hair loss)
14. Known hypersensitivity to any of the products to be administered during the study (such as JMT103)
15. Not suitable for this study as determined by the investigator due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage change of urinary N-terminal telopeptide of type 1 collagen/creatine (U-NTX/Cr) from baseline to week 13 | From enrollment to week 13.

SECONDARY OUTCOMES:
Incidence and type of adverse events (AEs) | From enrollment to 90 days after the last dose
Incidence of Skeletal-related event（SRE） | From enrollment to 90 days after the last dose
  SRE is defined as pathological fracture, radiotherapy to bone, surgery to bone, or spinal cord compression.
Change in Pain Score (Brief Pain Inventory-Short Form，BPI-SF) | From enrollment to 90 days after the last dose
Trough plasma concentration （Ctrough） | From enrollment to 90 days after the last dose
Percentage change in serum C-terminus peptide (of Type 1 Collagen) from baseline | From enrollment to 90 days after the last dose
Percentage change in serum bone-specific alkaline phosphatase (bALP) from baseline | From enrollment to 90 days after the last dose
Number of patients with anti-JMT103 antibodies | From enrollment to 90 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided